CLINICAL TRIAL: NCT00914251
Title: Positive Vascular Effect of Hesperidin in Subjects Affected by Metabolic Syndrome
Brief Title: Vascular Effects of Hesperidin in Metabolic Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Stefano Rizza, Medicine Internal Department
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 073/09
Record Dates: First submitted 2009-06-03; First posted 2009-06-04 (Estimated); Last update posted 2009-06-17 (Estimated); Status verified 2009-06

CONDITIONS: Endothelial Dysfunction; Metabolic Syndrome
Keywords: endothelial; metabolic syndrome; hesperidin
MeSH Terms: conditions — Metabolic Syndrome | interventions — Hesperidin

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Hesperidin, 500 mg per day (Active Comparator): 500 mg daily of oral Hesperidin for 3 weeks
  Interventions: Drug: Hesperidin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hesperidin — Administration of oral Hesperidin, 500 mg/daily
  Arms: Hesperidin, 500 mg per day
Drug: Placebo — Administration of oral Placebo, 500 mg/daily
  Arms: Placebo

SUMMARY:
It has been suggested that cardiovascular risk factors either independently or in cluster (metabolic syndrome) increase the risk of both type 2 diabetes (DM2) and cardiovascular diseases (CVD). Consumption of citrus fruits is linked to reduced cardiovascular morbidity and mortality. Hesperidin is a flavanone abundant in citrus fruit with putative vasodilator actions in vitro. While molecular mechanisms of vascular actions of hesperidin begin to be explored, no data on in vivo vascular effect of this flavanone has been ever acquired.

ELIGIBILITY:
Inclusion Criteria:

* Metabolic Syndrome (ATPIII criteria)
* BMI <35
* Age 20-55

Exclusion Criteria:

* History of cancer.
* History of cardiovascular diseases.
* Any other acute or chronic illness which requires administration of steroids or other drugs able to interfere with glucose or lipid metabolism.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-03 (Actual); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Safety of oral supplementation of hesperidin | 3 weeks

SECONDARY OUTCOMES:
Endothelial function assessed by FMD %. Inflammatory status assessed by biochemical markers. | 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rome Tor Vergata, Rome, Rome, Italy

REFERENCES:
- [Background] Muniyappa R, Hall G, Kolodziej TL, Karne RJ, Crandon SK, Quon MJ. Cocoa consumption for 2 wk enhances insulin-mediated vasodilatation without improving blood pressure or insulin resistance in essential hypertension. Am J Clin Nutr. 2008 Dec;88(6):1685-96. doi: 10.3945/ajcn.2008.26457. PMID 19064532
- [Background] Collins QF, Liu HY, Pi J, Liu Z, Quon MJ, Cao W. Epigallocatechin-3-gallate (EGCG), a green tea polyphenol, suppresses hepatic gluconeogenesis through 5'-AMP-activated protein kinase. J Biol Chem. 2007 Oct 12;282(41):30143-9. doi: 10.1074/jbc.M702390200. Epub 2007 Aug 27. PMID 17724029
- [Derived] Rizza S, Muniyappa R, Iantorno M, Kim JA, Chen H, Pullikotil P, Senese N, Tesauro M, Lauro D, Cardillo C, Quon MJ. Citrus polyphenol hesperidin stimulates production of nitric oxide in endothelial cells while improving endothelial function and reducing inflammatory markers in patients with metabolic syndrome. J Clin Endocrinol Metab. 2011 May;96(5):E782-92. doi: 10.1210/jc.2010-2879. Epub 2011 Feb 23. PMID 21346065